CLINICAL TRIAL: NCT00911157
Title: Clinical Evaluation of GSK576428 (Fondaparinux Sodium) in the Treatment of Acute Deep Vein Thrombosis (DVT)
Brief Title: The Treatment of Acute Deep Vein Thrombosis (DVT) of GSK576428 (Fondaparinux Sodium) in Japanese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111436
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2010-06-10 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Thrombosis, Venous
Keywords: Pulmonary thromboembolism; contrast-enhanced MDCT; Deep Vein Thrombosis; Fondaparinux sodium
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Fondaparinux; Heparin

ARMS (2):
- Fondaparinux (Experimental)
  Interventions: Drug: Fondaparinux sodium
- unfractionated heparin (Other)
  Interventions: Drug: unfractionated heparin (UFH)

INTERVENTIONS:
Drug: Fondaparinux sodium — The dose of Fondaparinux will be determined based on a subject's body weight (< 50 kg, 5 mg; 50 to 100 kg, 7.5 mg; >100 kg, 10 mg) and administered once daily by subcutaneous (SC) injection.
  Other Names: GSK576428
  Arms: Fondaparinux
Drug: unfractionated heparin (UFH) — UFH therapy will be started on Day 1 while adjusting activated partial thromboplastin time (aPTT) to maintain aPTT 1.5 to 2.5 times control.
  Arms: unfractionated heparin

SUMMARY:
The primary objective of this study is to evaluate the efficacy (as measured by the rate of recurrent symptomatic Venous Thromboembolism [VTE] (i.e., Pulmonary thromboembolism [PE] and Deep Vein Thrombosis [DVT])) and safety of GSK576428 as the initial treatment in subjects with acute symptomatic DVT in an open-label design.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acute proximal DVT based on contrast-enhanced Multi detector-row CT (MDCT) (not more than 10 days after the onset of the symptoms of DVT)
* Age:20 years
* Gender: No restriction
* Hospitalization status: Subjects who are able to stay at the hospital at least during the initial treatment period
* Written informed consent from the subject him/herself or his/her legally acceptable representative. Written informed consent from the subject's legally acceptable representative must be obtained if the subject is incapable of giving consent

Exclusion Criteria:

* Symptomatic PE
* Requirement for surgical thrombectomy, catheter intervention and thrombolytic therapy for the current DVT
* Subjects (for example, with free-floating thrombus in the femoral vein or ilium by MDCT at screening) for whom insertion of inferior vena cava filter is indicated or subjects in whom inferior vena cava filter is present
* Anticoagulant therapy for at least 24 hours to treat the current episode prior to entry into the study
* Active, clinically significant bleeding
* Thrombocytopenia (platelet count <10×10⁴/µL at screening)
* Concurrent conditions with bleeding risk (e.g., ulcer of the gastrointestinal tract, diverticulitis of the gastrointestinal tract, colitis, acute bacterial endocarditis, severe hypertension, or severe diabetes) or bleeding tendency
* Severe hepatic disorder
* Known hypersensitivity to heparin, low-molecular-weight heparin (LMWH) or warfarin
* Previous history of cerebral hemorrhage
* Brain, spinal, or ophthalmological surgery within 3 months prior to entry into this study
* Previous history of Heparin-induced thrombocytopenia
* Patients for whom anticoagulant therapy is contraindicated or who cannot be taken off anticoagulant therapy due to coexistent condition (e.g. prosthetic heart valve implant)
* Severe renal disorder (serum creatinine >2.0 mg/dL [180 µmol/L] at screening) in a well hydrated subject
* QT interval prolonged (QT interval corrected by Bazett's formula [QTcB] ≥450 msec; for patients with bundle branch block QTcB ≥480 msec) at screening
* Documented hypersensitivity to contrast media
* Use of any contraindicated drug that cannot be combined with the injection of contrast medium [e.g., antihyperglycemics, such as biguanides (metformin hydrochloride, buformin hydrochloride)]
* Participation in any other therapeutic drug study or a clinical study within 6 months prior to entry into this study
* Previous participation in a study of GSK576428 [Fondaparinux Sodium; including the studies of Org31540/SR90107A (ex-project code)] or previous exposure to the therapeutic dose of GSK576428
* Drug or alcohol abuse
* Systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg
* Recent surgery within 3 days prior to entry into the study
* Life expectancy <3 months
* Pregnant women, nursing mothers, women who may be pregnant, or women contemplating pregnancy during the study period
* Others whom the investigator or subinvestigator considers not eligible for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Japan (17):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Nakamura M, Okano Y, Minamiguchi H, Munemasa M, Sonoda M, Yamada N, Hanzawa K, Aoyagi N, Tsujimoto H, Sarai N, Nakajima H, Kunieda T. Multidetector-row computed tomography-based clinical assessment of fondaparinux for treatment of acute pulmonary embolism and acute deep vein thrombosis in Japanese patients. Circ J. 2011;75(6):1424-32. doi: 10.1253/circj.cj-10-1036. Epub 2011 Apr 22. PMID 21512258
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111436 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111436 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111436 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Fondaparinux Sodium (FPX): The dose of FPX was determined based on a participant's body weight (<50 kg, 5 mg; 50 to 100 kg, 7.5 mg; >100 kg, 10 mg) and was administered once daily by subcutaneous (SC) injection for 5-10 days as a general rule. Concomitant warfarin therapy (administered no later than 72 hours after the first dose of FPX) was continued up to Day 90 (±7) at a dose adjusted to maintain the prothrombin time international normalized ratio (PT-INR) between 1.5 and 3.0.
- Unfractionated Heparin (UFH): The dose of UFH was adjusted to maintain activated partial thromboplastin time (APTT) at 1.5-2.5 times control and was administered by intravenous (IV) drip bolus injection followed by IV infusion for 5-10 days as a general rule. Concomitant warfarin therapy (administered no later than 72 hours after the first dose of UFH) was continued up to Day 90 (±7) at a dose adjusted to maintain the PT-INR between 1.5 and 3.0.
Period: Overall Study
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Started | 29 | 10
Completed | 22 | 8
Not Completed | 7 | 2
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Need for prohibited drug (heparin) | 1 | 0
Not completed — Need to treat for lung cancer | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH) | Total
Number analyzed (Participants) | 28 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] — Full Analysis Set (FAS): 29 and 10 participants, respectively. One participant in each group whose data for the primary efficacy endpoint (contrast-enhanced MDCT) were missing were excluded.
  years | 64.5 (19.7) | 76.1 (12.2) | 67.3 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants] — FAS
  Participants
    Female | 15 | 9 | 24
    Male | 13 | 0 | 13
Race/Ethnicity, Customized [Number; unit: participants] — FAS
  participants
    Asian-Japanese | 28 | 9 | 37
Number of Participants with the Indicated Body Weight [Number; unit: participants] — Participants were weighed at Screening (within 10 days before randomization). FAS
  participants
    <50 kg | 8 | 3 | 11
    50-100 kg | 20 | 6 | 26
    >100 kg | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Recurrent or New Symptomatic Venous Thromboembolism (VTE)
Description: VTE (pulmonary thromboembolism [PE] and/or deep vein thrombosis [DVT]) was adjudicated blindly by the Central Independent Adjudication Committee of Efficacy (CIACE).
Time Frame: From Day 1 to Day 90 (±7 days)
Population: Full Analysis Set (FAS): all participants receiving at least one dose of medication (FPX or UFH) who had efficacy data and had a confirmed diagnosis of acute symptomatic deep vein thrombosis (DVT)
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 28 | 9
percentage of participants | 0 | 0

2. Secondary Outcome: Percentage of Participants With Recurrent or New Symptomatic/Asymptomatic VTE (by Type)
Description: VTE (pulmonary thromboembolism [PE] and/or deep vein thrombosis [DVT]) was adjudicated blindly by the CIACE.
Time Frame: From Day 1 to Day 90 (±7 days)
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 28 | 9
percentage of participants
  Symptomatic DVT only | 0 | 0
  (Symptomatic) Non-fatal PE | 0 | 0
  (Symptomatic) Fatal PE | 0 | 0
  Asymptomatic DVT only | 3.6 | 0
  Asymptomatic PE | 0 | 0

3. Secondary Outcome: Percentage of Participants With Perfusion Lung Scan Results Scored as Improved, no Change, or Worse Compared to Baseline
Description: Classifications of "Improved," "No change," or "Worse" were adjudicated blindly by the CIACE.
Time Frame: Baseline, single day between Day 5 and Day 10 (the day when the medication [FPX or UFH] was finished /discontinued) (±1 day)
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 28 | 9
percentage of participants
  Improved | 18.5 | 11.1
  No Change | 81.5 | 88.9
  Worse | 0 | 0

4. Secondary Outcome: Total Perfusion Score at Baseline and Mean Change From Baseline at Day 5-10
Description: Change from baseline was calculated as the score on the day medication was finished/discontinued (anywhere from Day 5 to Day 10) minus the baseline score. The perfusion score (0: no perfusion; 0.25, 0.5, 0.75, 1: normal) in each of the six lobes of the lung was adjudicated blindly by the CIACE. Total perfusion score (r) was calculated as: r = (0.25 x right lower lobe) + (0.12 x right middle lobe) + (0.18 x right upper lobe) + (0.20 x left lower lobe) + (0.12 x lingula) + (0.13 x left upper lobe).
Time Frame: as for outcome 3
Population: FAS
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 28 | 9
points on a scale
  Baseline | 0.944 (0.087) | 0.959 (0.048)
  Change from Baseline | 0.015 (0.034) | 0.004 (0.011)

5. Secondary Outcome: Percentage of Participants With a Bleeding Event
Description: Bleeding events (major bleeding [clinically overt bleeding with fatality, location in a critical organ, a fall in hemoglobin >=2 grams (g)/deciliter (dL), or a transfusion >=2 units]; minor bleeding [clinically overt bleeding and not adjudicated as major bleeding], and no bleeding) were adjudicated blindly by the Central Independent Adjudication Committee of Safety (CIACS).
Time Frame: Initial treatment period (from the first dose of FPX/UFH to N days after the last dose of FPX/UFH; specified based on creatinine clearance [CLcr]; N=3, CLcr >=50 mL/min; N=4, 30 =< CLcr < 50 mL/min; N=9, CLcr < 30 mL/min).
Population: Safety Population: all participants who received at least one dose of medication (FPX or UFH).
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 29 | 10
percentage of participants
  Major bleeding | 3.4 | 0
  Minor bleeding only | 3.4 | 0
  Any bleeding (major and/or minor bleedings) | 6.9 | 0

ADVERSE EVENTS:
Time Frame: SAEs and AEs were evaluated during the initial treatment period (from the first dose of FPX/UFH to N days after the last dose of FPX/UFH; specified based on creatinine clearance [CLcr].
Description: SAEs, serious adverse events; AEs, adverse events. CLcr was determined at the last dose of FPX/UFH; N=3, CLcr >=50 mL/min; N=4, 30 =< CLcr < 50 mL/min; N=9, CLcr < 30 mL/min). CLcr was calculated according to the Cockcroft and Gault formula: CLcr = (140 - age) × weight (kilograms)/(72 × serum creatinine [mg/dL]) × 0.85 (in case of women).
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Serious Adverse Events (participants affected / at risk) | 1/29 | 1/10
Other Adverse Events (participants affected / at risk) | 18/29 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux Sodium (FPX) (N=29) | Unfractionated Heparin (UFH) (N=10)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux Sodium (FPX) (N=29) | Unfractionated Heparin (UFH) (N=10)
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 0 | 1
Coagulation time prolonged (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Injection site haemorrhage (General disorders) | 1 | 0
Xerosis (General disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.